CLINICAL TRIAL: NCT01993121
Title: Exercise and Type 2 Diabetes: Gender and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 02-0514
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; exercise; heart; cardiovascular
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Three-month exercise training program (Experimental): All subjects will perform three months of supervised exercise training.
  Interventions: Other: Supervised Exercise Training

INTERVENTIONS:
Other: Supervised Exercise Training — All subjects will perform three months of supervised exercise training.

SUMMARY:
The objective of the current proposal is to evaluate the importance of blood vessel dysfunction and heart dysfunction to overall exercise impairments in type 2 diabetes and their contribution to the gender differences observed in exercise capacity. Importantly, treatments that improve blood vessel function in persons with type 2 diabetes can be used to directly assess whether impairment in blood vessel function and ultimately exercise performance, can be improved and whether the degree of improvement differs between the sexes.

Hypothesis 1. Uncomplicated type 2 diabetes more adversely affects exercise capacity in women than men.

Hypothesis 2. Blood vessel function and cardiac function are more significantly impaired in women with type 2 diabetes than men and contribute to the gender differences in exercise capacity.

Hypothesis 3. Restoration of blood vessel function will improve exercise capacity more in women than men with type 2 diabetes.

DETAILED DESCRIPTION:
Subjects will come in for a total of seven research visits. Four initial study visits before exercise training for three months and then subjects will repeat the testing.

1. Initial exam. A history and physical exam will be performed. Blood will be drawn for measurements of overall health. Resting electrocardiogram will be obtained. The Low Level Physical Activity Recall (LOPAR) questionnaire will be administered.
2. Dual Energy X-ray Absorptiometry (DEXA) will be carried out during visit two. A familiarization bicycle ergometer test will also be performed on this day.
3. During visit three, a euglycemic clamp will be performed.
4. During visit four, echocardiographic measurements will be made and a diet interview will be performed.
5. On visit five, measures of blood vessel-dependent vasodilation will be performed. Repeated brachial artery diameter and forearm blood flow responses to cuff occlusion will be measured separately on this occasion.
6. On visit six, arterial stiffness will be measured. Subjects will also perform a graded bicycle exercise test.
7. On visit seven, subjects will perform constant level bicycle tests.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 30 and 55 years
* Persons with type 2 diabetes taking only certain oral medications (
* Pre-menopausal women
* Persons with type 2 diabetes who have a total HbA1c level <9%
* Persons with a BMI between 25-35.

Exclusion Criteria:

* Current smokers or anyone who has smoked within the last year
* Persons who have clinically evident distal symmetrical neuropathy
* Abnormal lipid levels (total cholesterol >200, LDL-cholesterol level >130, or triglyceride level >250).
* Persons with regional wall motion abnormalities, left ventricular wall thickness >1.1 cm , or decreased contractility.
* Persons will also be excluded if they have evidence of ischemic heart disease by history or abnormal resting or exercise electrocardiogram (ECG).
* Presence of systolic blood pressure >140 mmHg at rest or >250 mmHg with exercise or diastolic pressure >90 mmHg at rest or >105 mmHg with exercise will be grounds for exclusion.
* Subjects will be excluded who have peripheral arterial disease.
* Persons with autonomic insufficiency, assessed by measuring variation in RR intervals with cycled breathing and by presence of a >20 mm fall in upright blood pressure without a change in heart rate, will be excluded.
* Subjects with proteinuria (urine protein >200 mg/dl) or a creatinine > 2 mg/dl, suggestive of renal disease will be excluded.
* Controls will not be accepted with an immediate family history of Type 2 Diabetes Mellitis

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in cardiovascular exercise performance | baseline and 3 months
  Subjects' peak oxygen consumption will be tested on a stationary bike before and after 3 months of exercise training.
Changes from baseline in cardiovascular exercise performance | baseline and 3 months
  Subjects' oxygen uptake kinetics will be tested on a stationary bike before and after 3 months of exercise training.
Changes from baseline in cardiovascular exercise performance | baseline and 3 months
  Subjects' tissue oxygen saturation will be tested during exercise testing before and after 3 months of exercise training.

SECONDARY OUTCOMES:
Changes from baseline in endothelial function will be measured | baseline and 3 months
  Endothelial-dependent vasodilation will be determined in the peripheral circulation by measurement of changes in brachial artery diameter in response to cuff occlusion.
Changes from baseline in endothelial function will be measured | baseline and 3 months
  Forearm blood flow will be assessed by plethysmography before and after cuff occlusion.
Changes from baseline in diastolic function will be measured | baseline and 3 months
  The role of diastolic function in the exercise impairments will be examined using advanced echocardiographic techniques during rest and exercise

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Regensteiner, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States